CLINICAL TRIAL: NCT05092698
Title: The Efficacy of Vitamin D Supplementation in Patients With Severe and Extremely Severe COVID-19
Acronym: COVID-VIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-VIT
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV2 Infection
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV2); coronavirus disease 2019 (COVID-19); severe and extremely severe disease; Vitamin D; cholecalciferol
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vit_D_suppl (Active Comparator): Patients will receive 60,000 IU of cholecalciferol dissolved in 45 ml herbal oil orally or via feeding tube weekly followed by 5,000 IU of cholecalciferol (two drops) daily until discharge or death.
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)
- Vit_D_placebo (Placebo Comparator): Patients will receive 45 ml of herbal oil orally or via feeding tube followed by 45 ml of herbal oil weekly followed by two drops of herbal oil daily until discharge or death.
  Interventions: Dietary Supplement: Herbal oil

INTERVENTIONS:
Dietary Supplement: Vitamin D (cholecalciferol) — Patients will receive 60,000 IU of cholecalciferol dissolved in 45 ml herbal oil orally or via feeding tube after serum Vitamin D concentrations measurement followed by the same dose of cholecalciferol weekly and 5,000 IU of cholecalciferol (two drops) daily until discharge or death.
  Arms: Vit_D_suppl
Dietary Supplement: Herbal oil — Patients will receive 45 ml of herbal oil orally or via feeding tube after serum Vitamin D concentrations measurement followed by the same dose of pure herbal oil weekly and two drops of herbal oil daily until discharge or death.
  Other Names: Placebo
  Arms: Vit_D_placebo

SUMMARY:
Despite the successful treatment of patients with moderate coronavirus disease 2019 (COVID-19), outcomes for patients with severe disease remain unsatisfactory. In this category of patients, the course of the disease is complicated by the development of acute respiratory distress syndrome (ARDS) and the need for mechanical ventilation in the intensive care unit (ICU). Mortality in this category of patients reaches 85%. The lack of effective treatment for COVID-19 has prompted scientists to look for new strategies to reduce the incidence and severity of COVID-19, disease progression, and mortality.

Disease severity and mortality rates due to COVID-19 infection are greater in the elderly and chronically ill patients, populations at high risk for vitamin D deficiency. Vitamin D plays an important role in immune function and inflammation.

A number of experimental studies have shown that stimulation of vitamin D receptors can improve the course of ARDS due to inhibition of the hyperimmune inflammatory response, regulation of the renin-angiotensin system, modulation of neutrophil activity, maintenance of the integrity of the pulmonary epithelial barrier and stimulation of epithelial repair, as well as by reducing hypercoagulation.

Several studies on ICU patients have reported that low vitamin D (25(OH)D) concentrations are associated with a higher risk of negative outcomes such as death, organ failure, prolonged mechanical ventilation, a higher rate of ventilation-associated pneumonia, and sepsis.

While the available evidence to-date, from largely poor-quality observational studies, may be viewed as showing a trend for an association between low serum 25(OH)D levels and COVID-19 related health outcomes, this relationship was not found to be statistically significant. Calcifediol supplementation may have a protective effect on COVID-19 related ICU admissions.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy of vitamin D (cholecalciferol) supplementation in patients with severe and extremely severe disease caused by the SARS-CoV-2 virus, admitted to an ICU of the COVID-center on the first day and in dynamics until discharge from the hospital or death. Patients with vitamin D deficiency [25-hydroxyvitamin D (25(OH)D) ≤ 30 ng/ml] will be randomized to two groups: 1 - patients will receive 60,000 IU of cholecalciferol supplementation; 2 - patients will receive matched placebo.

The demographic and clinical data will be collected. Laboratory data (hemoglobin, lymphocytes, neutrophil to lymphocyte ratio, D-dimer level, Interleukin-6, procalcitonin, ferritin, glucose level, high-sensitive troponin Т, vitamin D level (25(OH)D), acid-base balance, signs of a secondary bacterial infection, immunogram, Von Willebrand factor antigen and Instrumental data (CT-scan, Electrocardiography, echocardiography, arterial and venous ultrasound investigation) will be analysed. The frequency of complications, duration of mechanical ventilation, length of stay in the ICU and in the hospital, and mortality will be evaluated.

This study is single-centre prospective randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* all patients with COVID-19 admitted to the ICU with vitamin D deficiency [25-hydroxyvitamin D (25(OH)D) ≤ 30 ng/ml]

Exclusion Criteria:

* less than 24 hours in ICU by any reason
* chronic decompensated disease with extrapulmonary organ dysfunction (tumour progression, liver cirrhosis, congestive heart failure) with a life expectancy of less than 48 hours
* atonic coma
* allergic reaction on cholecalciferol or herbal oil

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Сomplete blood count | Change from baseline on day 5 during ICU treatment
  Сomplete blood count
Сomplete blood count dynamics 1 | Change from baseline on day 10 during ICU treatment
  Сomplete blood count
Сomplete blood count dynamics 2 | Change from baseline on day 15 during ICU treatment
  Сomplete blood count
Сomplete blood count dynamics 3 | Change from baseline on day 21 during ICU treatment
  Сomplete blood count
C-reactive protein | Change from baseline on day 5 during ICU treatment
  Concentration of C-reactive protein
C-reactive protein 1 | Change from baseline on day 10 during ICU treatment
  Concentration of C-reactive protein
C-reactive protein 2 | Change from baseline on day 15 during ICU treatment
  Concentration of C-reactive protein
C-reactive protein 3 | Change from baseline on day 21 during ICU treatment
  Concentration of C-reactive protein
Von Willebrand factor antigen | Change from baseline on day 7 during ICU treatment
  Concentration of Von Willebrand factor antigen
Thrombotic complications | 60 days
  Arterial or venous thrombotic complications
Immunogram | Change from baseline on day 7 during ICU treatment
  The amount of NKT cells (CD3+CD56+CD16+), NK cells (CD3-CD56+CD16+)
Proinflammatory marker | Change from baseline on day 5 during ICU treatment
  Concentration of D-dimer
Proinflammatory marker 1 | on day 10 during ICU treatment
  Concentration of D-dimer
Proinflammatory marker 2 | on day 15 during ICU treatment
  Concentration of D-dimer
Proinflammatory marker 3 | on day 21 during ICU treatment
  Concentration of D-dimer
inflammatory marker | Change from baseline on day 5 during ICU treatment
  Concentration of Interleukin-6
inflammatory marker 1 | Change from baseline on day 10 during ICU treatment
  Concentration of Interleukin-6
inflammatory marker 2 | Change from baseline on day 15 during ICU treatment
  Concentration of Interleukin-6
inflammatory marker 3 | Change from baseline on day 21 during ICU treatment
  Concentration of Interleukin-6
Infection marker | Change from baseline on day 5 during ICU treatment
  Concentration of Procalcitonin
Infection marker 1 | Change from baseline on day 10 during ICU treatment
  Concentration of Procalcitonin

SECONDARY OUTCOMES:
Mortality | 60 days
  The dead and survived patients ratio
Mechanical ventilation duration | 30 days
  The amount of mechanical ventilation days
Non-invasive Mechanical ventilation duration | 30 days
  The amount of Non-invasive mechanical ventilation days
Length of stay in the ICU | 60 days
  The amount of day of ICU treatment
Length of stay in the hospital | 60 days
  The amount of day of hospital treatment
Infection complications | 60 day
  The amount of Infection complications

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana V Klypa, ScD, Study Chair — Federal Research Clinical Center of Federal Medical & Biological Agency
Locations (1):
- Federal Research Clinical Center of Federal Medical & Biological Agency, Moscow, Russia

REFERENCES:
- [Background] Bassatne A, Basbous M, Chakhtoura M, El Zein O, Rahme M, El-Hajj Fuleihan G. The link between COVID-19 and VItamin D (VIVID): A systematic review and meta-analysis. Metabolism. 2021 Jun;119:154753. doi: 10.1016/j.metabol.2021.154753. Epub 2021 Mar 24. PMID 33774074
- [Background] Bychinin MV, Klypa TV, Mandel IA, Andreichenko SA, Baklaushev VP, Yusubalieva GM, Kolyshkina NA, Troitsky AV. Low Circulating Vitamin D in Intensive Care Unit-Admitted COVID-19 Patients as a Predictor of Negative Outcomes. J Nutr. 2021 Aug 7;151(8):2199-2205. doi: 10.1093/jn/nxab107. PMID 33982128
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Kong J, Zhu X, Shi Y, Liu T, Chen Y, Bhan I, Zhao Q, Thadhani R, Li YC. VDR attenuates acute lung injury by blocking Ang-2-Tie-2 pathway and renin-angiotensin system. Mol Endocrinol. 2013 Dec;27(12):2116-25. doi: 10.1210/me.2013-1146. Epub 2013 Nov 6. PMID 24196349
- [Derived] Bychinin MV, Klypa TV, Mandel IA, Yusubalieva GM, Baklaushev VP, Kolyshkina NA, Troitsky AV. Effect of vitamin D3 supplementation on cellular immunity and inflammatory markers in COVID-19 patients admitted to the ICU. Sci Rep. 2022 Nov 3;12(1):18604. doi: 10.1038/s41598-022-22045-y. PMID 36329227